CLINICAL TRIAL: NCT05742360
Title: Effect of CPAP on 24-Hour Blood Pressure in the Excessively Sleepy Obstructive Sleep Apnea Subtype
Brief Title: Effect of CPAP on Blood Pressure in Excessively Sleepy Obstructive Sleep Apnea Subtype
Status: Recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Ulysses Magalang MD, Professor of Internal Medicine, Ohio State University
Other Study IDs: 2022H0323
Record Dates: First submitted 2023-01-26; First posted 2023-02-24 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Obstructive Sleep Apnea
Keywords: Excessively Sleepy Symptom Subtype
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The blood samples will be used to determine levels of BP medications and serum creatinine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- OSA subjects with the excessively sleepy symptom subtype treated with CPAP: Patients with the excessively sleepy symptom subtype who accept CPAP therapy
  Interventions: Device: CPAP therapy

INTERVENTIONS:
Device: CPAP therapy — CPAP treatment of obstructive sleep apnea with the excessively sleepy symptom subtype

SUMMARY:
The primary objective of this study is to determine the longer-term (6 months) effect of CPAP therapy on change in 24-hour mean blood pressure (24hMBP) in OSA subjects with the excessively sleepy symptom subtype.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, observational, two-center study involving newly diagnosed subjects with moderate-severe OSA with the excessively sleepy symptom subtype.

Variables of Interest: Change in 24-hour ambulatory BP, change in sitting BP, change in reaction time by psychomotor vigilance test (PVT)

Participants will complete questionnaires that pertain to demographics, lifestyle factors, and co-morbidities. The blood samples will be used to determine levels of BP medications and serum creatinine. Measurements will be collected at baseline and at 6-month follow-up visits.

Data Analysis Approach: To correct for potential bias in the non-randomized comparison, the investigators will apply a Propensity Score (PS) Design via subclassification. Models to derive the PS values used in this design will include a number of covariates relevant to CPAP adherence, including age, sex, obesity (BMI, neck circumference, waist-to-hip ratio), current smoking, history of hypertension, diabetes mellitus (history, medications), lipid profile, hyperlipidemia (history, medications), family history of premature coronary disease, Charlson comorbidity index, physical activity (IPAQ), diet, OSA severity (AHI, ODI4, T90), sleepiness (Epworth Sleepiness Scale), educational attainment, socioeconomic status (postcode), insomnia symptoms (Insomnia Symptom Questionnaire), anxiety and depression-related symptoms (Patient Health Questionnaire-2), self-efficacy (General self-efficacy scale), and medication adherence (Medication Adherence Report Scale [MARS-5]). Baseline values of outcome measures will also be included in the PS model. After creating the PS design, all analyses are performed accounting for PS subclass as a categorical stratification factor. Evaluations of the CPAP effect on binary outcomes are performed utilizing conditional logistic regression. Similarly, CPAP effects in the context of survival analyses (e.g., Cox Proportional Hazards models) or on continuous outcomes (e.g., linear regression) are assessed by including PS subclass as a categorical covariate in all models.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Moderate-severe OSA (defined as ODI ≥10 events/hour) via Polysomnography (PSG) or Home Sleep Apnea Study (HSAT) done based on clinical grounds
* Excessively sleepy subtype determined by patient-reported symptoms
* Willing to accept CPAP therapy
* An elevated baseline office BP defined as ≥120 or ≥80 mmHg
* Planned PAP (CPAP or bi-level PAP) treatment by treating provider

Exclusion Criteria:

* Recent changes (within 3 months) to BP medications among those who are on these medications
* Unable to apply ABPM cuff
* Current use of CPAP or other OSA treatments
* Resting, awake SaO2 <90% or use of home oxygen therapy
* New York Heart Association (NYHA) categories III-IV of heart failure
* Presence of Cheyne-Stokes Respiration (CSR) in sleep study identified by typical crescendo-decrescendo pattern of respiration with associated apneas and/or hypopneas in the absence of inspiratory flow limitation
* Predominantly central sleep apnea (AHI≥15 events/hour, with >50% central events [apnea or hypopnea])
* Life expectancy <2 years
* Pregnancy
* Clinical history of chronic kidney disease (Stage 5) requiring dialysis, or renal transplant
* Systolic BP > 180 mmHg

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults between the ages of 18 to 75 years old with moderate-severe obstructive sleep apnea (OSA) with excessively sleepy symptom subtype. OSA diagnosis will be defined as an apnea/hypopnea index (AHI) >or =5 episodes per hour.
Sampling Method: Probability Sample
Enrollment: 227 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in 24-hour Mean Blood Pressure | Change from baseline 24-hour Mean Blood Pressure at 6-months after initiation of CPAP therapy
  24-hour Mean Blood Pressure obtained from ambulatory blood pressure monitoring (ABPM)

SECONDARY OUTCOMES:
Nocturnal Mean BP | Change from baseline nocturnal Mean Blood Pressure at 6-months after initiation of CPAP therapy
  Nocturnal Mean Blood Pressure obtained from ambulatory blood pressure monitoring (ABPM)
Reciprocal of Reaction Time | Change from baseline reaction time at 6-months after initiation of CPAP therapy
  Reciprocal of reaction time obtained by Psychomotor Vigilance Test

CONTACTS AND LOCATIONS:
Overall Officials: Ulysses Magalang, MD, Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - The Ohio State University - Martha Morehouse Medical Pavilion, Suite 2600, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No